CLINICAL TRIAL: NCT04568707
Title: Evaluation of Biological Response to SARS-COV2 in Patients With Pre-existing Neurological Disease or With New Neurological Manifestations of COVID-19
Brief Title: Evaluation of Biological Response to SARS-COV2 (COVID-19) in Patients With Pre-existing Neurological Disease or Newly Neurological Symptoms (BIO-COCO-NEUROSCIENCES)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Paris Brain Institute (ICM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP200845
Record Dates: First submitted 2020-08-31; First posted 2020-09-29 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Covid19; Neurologic Manifestations; Psychiatric Manifestations
Keywords: COVID-19; neurological disease; Multiple Sclerosis; psychiatric disease; biology,; biocollection,; biomarkers,; DNA,; Parkinson's Disease
MeSH Terms: conditions — COVID-19; Neurologic Manifestations; Nervous System Diseases; Multiple Sclerosis; Mental Disorders; Parkinson Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Covid-19 infection (Experimental): Covid-19 infection defined by a positive PCR or a typical chest scanner of Covid-19 infection or a positive serology or a typical clinical picture in a pandemic period
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — blood sample for serum (serology, biomarkers) and DNA

SUMMARY:
Patients with neurological or psychiatric symptoms or pre-existing disease will be sampled (blood for serum and DNA or saliva for DNA) at inclusion and at M6 (blood) and M12 (blood) depending on their pathology. Sampling will be done either at hospital if patient is on site for routine care or at home if no consultation is scheduled at hospital.

ELIGIBILITY:
1. Age over 18 yo
2. Patient having presented or presenting a Covid-19 infection defined by a positive PCR or a typical chest scanner of Covid-19 infection or a positive serology or a typical clinical picture in a pandemic period
3. And patient with:

   1. a neurological or psychiatric manifestation de novo during or after the Covid-19 infection and/or
   2. either a chronic neurological or psychiatric pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
dosage of seric markers (anti-SARS-CoV2 IgG) or genetic markers (genetic variants) observed during COVID 19 infection in patients | 12 months
  dosage of seric markers (anti-SARS-CoV2 IgG) or genetic markers (genetic variants) observed during COVID 19 infection in patients

SECONDARY OUTCOMES:
Serum neurofilaments | 12 months
  Neurodegenerative markers (e.g., neurofilaments) associated with a neurological or psychiatric manifestation of Covid-19 infection

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié Salpétrière, Paris, France

REFERENCES:
- [Derived] Louapre C, Ibrahim M, Maillart E, Abdi B, Papeix C, Stankoff B, Dubessy AL, Bensa-Koscher C, Creange A, Chamekh Z, Lubetzki C, Marcelin AG, Corvol JC, Pourcher V; COVISEP and Bio-coco-neuroscience study group. Anti-CD20 therapies decrease humoral immune response to SARS-CoV-2 in patients with multiple sclerosis or neuromyelitis optica spectrum disorders. J Neurol Neurosurg Psychiatry. 2022 Jan;93(1):24-31. doi: 10.1136/jnnp-2021-326904. Epub 2021 Aug 2. PMID 34341142